CLINICAL TRIAL: NCT02738164
Title: Validation of the SEPSIS-3 Criterion for Sepsis and Septic Shock in the Emergency Department
Brief Title: SEPSIS 3 Critera for Risk Stratification in Emergency Patients
Acronym: SCREEN
Status: Completed | Type: Observational
Sponsor: Societe Française de Medecine d'urgence (Other)
Responsible Party: Sponsor
Other Study IDs: SCREEN_SFMU
Record Dates: First submitted 2016-04-02; First posted 2016-04-14 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Sepsis; Emergency
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators aim to evaluate the SEPSIS 3 criterion for "sepsis" and "septic shock" in a prospective manner.

Investigators will evaluate qSOFA performances and other SEPSIS 3 criterion in a population of emergency patients with infection

ELIGIBILITY:
Inclusion Criteria:

* Adult that present to the emergency department
* Diagnosis of infection by the treating emergency physician

Exclusion Criteria:

* Refuse to participate
* pregnancy
* prisoner
* Low acuity infection (localised, not requiring general treatment, without any abnormal vital parameters)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency patients with infection
Sampling Method: Non-Probability Sample
Enrollment: 879 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
In hospital mortality | 30 days

SECONDARY OUTCOMES:
admission in ICU | 30 days
length of ICU stay more than 72 hours | 30 days
Length of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, MD, PhD, Principal Investigator — SFMU
Locations (27):
- St Luc, Brussels, Belgium
- France (24):
  - CHU Angers, Angers
  - CHIPO, Beaumont S Oise
  - Avicenne, Bobigny
  - Saint Camille, Bry-sur-Marne
  - Dijon, Dijon
  - Grenoble, Grenoble
  - Longjumeau, Longjumeau
  - Lyon, Lyon
  - Princess Grace, Monaco
  - Nancy, Nancy
  - Nice, Nice
  - Ambroise Paré, Paris
  - Bichat, Paris
  - Cochin, Paris
  - HEGP, Paris
  - Lariboisière, Paris
  - Pitie-salpetriere, Paris
  - Saint-Antoine, Paris
  - St Louis, Paris
  - Tenon, Paris
  - Strasbourg, Strasbourg
  - Toulouse, Toulouse
  - Tours, Tours
  - Vienne, Vienne
- Clinic hospital Barcelona, Barcelona, Spain
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freund Y, Lemachatti N, Krastinova E, Van Laer M, Claessens YE, Avondo A, Occelli C, Feral-Pierssens AL, Truchot J, Ortega M, Carneiro B, Pernet J, Claret PG, Dami F, Bloom B, Riou B, Beaune S; French Society of Emergency Medicine Collaborators Group. Prognostic Accuracy of Sepsis-3 Criteria for In-Hospital Mortality Among Patients With Suspected Infection Presenting to the Emergency Department. JAMA. 2017 Jan 17;317(3):301-308. doi: 10.1001/jama.2016.20329. PMID 28114554